CLINICAL TRIAL: NCT05140551
Title: Investigating the Care That People With Diabetes Receive for Their Emotional Wellbeing
Brief Title: Emotional Wellbeing in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 301444
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes; Depression; Anxiety; Distress, Emotional; Diabetes Distress; Loneliness; Social Functioning; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Depression; Anxiety Disorders; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMPASS (Experimental): This is a single arm study. We are investigating COMPASS digital CBT.
  Interventions: Device: COMPASS: digital CBT

INTERVENTIONS:
Device: COMPASS: digital CBT — COMPASS is an evidence based digital CBT intervention with guided therapist support, tailored to treat anxiety and/or depression in long term conditions (LTCs). The intervention consists of eleven modules/sessions in which CBT techniques are taught. Users of COMPASS receive guided therapist support from a trained therapist. The guided support aims to help patients identify and apply the CBT skills outlined in COMPASS to meet their individual needs and experiences of living with LTC(s). The support can occur through in-site messaging or via the telephone.
  Other Names: COMPASS: Navigating your long-term condition

SUMMARY:
The investigators want to understand the feasibility and acceptability of implementing COMPASS: Online Cognitive behavioural therapy (CBT) in routine NHS care for individuals with diabetes. People with type 1 or type 2 diabetes with co-morbid psychological distress will be invited to take part in a pre-post implementation study of COMPASS: Online CBT for managing depression and anxiety in context of Long-Term conditions (LTCs). Patients with diabetes who are also experiencing depression and/or anxiety and/or diabetes specific distress will be recruited from: Improving Access to Psychological therapies (IAPT) services or clinics within Guys and St Thomas National Health Service (NHS) trust (GSTT) in London, United Kingdom (UK).

ELIGIBILITY:
IAPT (primary care recruitment)

Patients will be eligible for inclusion if they are:

* Adults aged 18 or above.
* Diagnosed with T1 diabetes or T2 diabetes
* Have been self-referred/been referred to Southwark or Hackney (London) IAPT service for psychological support.
* Speak English to a sufficiently high standard to allow them to interact with COMPASS.
* Have access to the internet.

GSTT (Secondary care recruitment)

The same criteria will be applied as above but with the additional criteria in place:

* Have psychological distress levels below the cut offs outlined by the service for face-to-face psychological treatment (see below for criteria):
* (Diabetes Distress Scale (DDS-17) mean score <4

and/or

- Patient Health Questionnaire (PHQ-9) score <19

and/or

- Generalised Anxiety Disorder Scale (GAD-7 score) <15

AND

- Diabetes Eating Problems Scale- Revised (DEPS-R) score <20)

or

- Are deemed eligible for digital support by a clinician for patients who have not been assessed using mental health screening tools.

IAPT (primary care recruitment)

The following exclusion criteria will be applied:

* Currently in receipt of psychological treatment for anxiety and/or depression.
* Evidence of a severe mental health disorder (including bipolar disorder or psychosis) and/or alcohol and/or drug dependency identified by highly trained IAPT therapists as part of routine care.
* Acute suicidal risk requiring a level of support that cannot be provided by therapists who are supporting patients remotely in their use of digital health interventions.

GSTT (secondary care recruitment)

As above but with the additional exclusion criteria below:

- Evidence of a diabetes related eating disorder requiring a level of support that cannot be provided by therapists who are supporting patients remotely in their use of digital health interventions evidenced through a DEPS-R score of ≥20.

Eligibility criteria for the qualitative study - Qualitative Patient and healthcare professionals (HCP) interviews:

* The investigators will interview participants who have experience of receiving COMPASS and those who do not uptake COMPASS.
* The investigators also aim to interview participants who commenced COMPASS and subsequently dropped out of treatment.
* The investigators will interview HCPs who have assessed and triaged patients for treatment, and those who have provided psychological support to individuals with diabetes.
* Patients and HCPs will be purposively sampled to achieve a mix of age, gender, ethnicity, clinical variables and/or professional experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
To assess the socio-demographic and clinical reach of COMPASS. | To be collected throughout the study duration (the study will run for an average of 12 months).
  Descriptive data, specifically frequencies documenting the number of individuals who are willing to use COMPASS, reasons documented for ineligibility/non-uptake and the sociodemographic and clinical profile of users vs non-users of COMPASS.
To assess the socio-demographic and clinical reach of COMPASS. | To be collected throughout the study duration (the study will run for an average of 12 months).
  Descriptive data on the types of treatment individuals with diabetes received throughout the study.
To assess the socio-demographic and clinical reach of COMPASS. | To be collected throughout the study duration (the study will run for an average of 12 months).
  Descriptive data documenting the number of individuals who consent to be contacted about research and subsequently give informed consent. The investigators will also report reasons for non-consent where this is disclosed.
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported mental health outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - General psychological distress: Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS)
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported mental health outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Depression: Patient health Questionnaire -9 (PHQ-9).
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported mental health outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Anxiety: Generalised anxiety disorder assessment-7 (GAD-7)
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported mental health outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Diabetes distress: Diabetes distress scale -17 (DDS-17)
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported psychosocial outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Loneliness: The revised University of California Los Angeles Loneliness scale (UCLA-R)
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported psychosocial outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Social Functioning: The Work and Social Adjustment Scale (WSAS)
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported psychosocial outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Health Related Quality of Life: The European Quality of Life scale (EQ-5D-3L)
To explore the potential efficacy of COMPASS by examining pre-post change scores on self-reported physical health outcomes (listed below). | To be collected at baseline, 12 weeks and 6 month follow up.
  - Glycaemic control: self-reported HbA1c levels.
To examine barriers and facilitators to the adoption of COMPASS from the perspective of both staff and patients. | To be collected at 12 weeks.
  Semi-structured interviews will be conducted to explore patient and health care professional (HCP) perceptions of the barriers and facilitators of using COMPASS in the context of diabetes.
To examine: i) number of patients who require digital support to use COMPASS ii) monthly referrals to COMPASS by staff. | To be collected at 12 weeks.
  The investigators will use descriptive statistics to quantify the number of patients who require digital support to use COMPASS and ii) monthly referrals to COMPASS by staff.
To assess the implementation of COMPASS in terms of patient adherence to COMPASS online sessions and number and duration of therapist support calls attended. | To be collected throughout the study duration (the study will run for an average of 12 months).
  Descriptive data on number of online sessions completed and number and duration of therapist support calls attended will be extracted from the COMPASS program.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Guys Hospital, London, Other
  - Emma Jenkinson, London
  - King's College London, London
  - South London and Maudsley, London

IPD SHARING:
Plan to Share IPD: No